CLINICAL TRIAL: NCT04064086
Title: A Patient-centered, System-based Approach to Improve Informed Dialysis Choice and Outcomes in Veterans With CKD
Brief Title: Trial to Evaluate and Assess the Effect of Comprehensive Pre-ESKD Education on Home Dialysis Use in Veterans
Acronym: TEACH-VET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-202; I01HX002639 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Hemodialysis; Peritoneal Dialysis
Keywords: Chronic kidney disease; Pre-dialysis education; Kidney Disease Education; Patient Education; Decision Making
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study compares a comprehensive education with the standard of care. Thus it is not possible to mask investigator, participant or care provider. However, our statistician will assess the outcomes aggregates in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comprehensive Pre-ESRD Patient Education (CPE) (Active Comparator): These patients will receive CPE for a total of up to 3 session in an intent-to-teach format, either via Face-to-face or telemedicine delivery.
  Interventions: Other: Comprehensive Pre-ESRD Patient Education (CPE)
- Enhanced Usual Care (Active Comparator): This group will receive usual care. This care will be enhanced by providing them with the freely available education material for the Kidney Disease Education
  Interventions: Other: Provision of the freely available resources for Kidney Disease Education

INTERVENTIONS:
Other: Comprehensive Pre-ESRD Patient Education (CPE) — Structured education session/s
  Other Names: Kidney Disease Education, CKD education, dialysis education
  Arms: Comprehensive Pre-ESRD Patient Education (CPE)
Other: Provision of the freely available resources for Kidney Disease Education — freely available resources
  Other Names: information brochure
  Arms: Enhanced Usual Care

SUMMARY:
This study is intended to correct an important systemic deficit in the care of chronic kidney disease (CKD), VHA's fourth most common healthcare condition with high mortality and healthcare burden. Currently, many Veterans with CKD have poor awareness of their condition. This leads to suboptimal care. The investigators anticipate that the proposed comprehensive pre-end stage renal disease (ESRD) education (CPE) will enhance Veterans' CKD knowledge and their confidence in making an informed selection of an appropriate dialysis modality, and lead to an increase in the use of home dialysis (HoD) - an evidence-based, yet underutilized dialysis modality. Further, this study will allow us to examine whether such Veteran-informed dialysis choice can improve Veteran and health services outcomes. If successful, this study may deliver a ready to roll-out strategy to meet the CKD care needs of the Veterans and reduce VHA healthcare costs.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is the 4th most common diagnosis among Veterans. Each year, over 13,000 Veterans transition from CKD to end stage renal disease (ESRD), a disease with high mortality and poor health related quality of life (HRQoL). Over 52,000 Veterans with ESRD are currently on dialysis and CKD/ESRD care costs VA over $18 billion per year. The majority of Veterans progressing from CKD to ESRD have limited to no awareness of CKD and its treatment options. This hinders Veterans' informed dialysis selection resulting in a gross underuse (7%) of home dialysis (HoD). As there are no significant differences in mortality among different dialysis modalities, VHA National Kidney Program and professional renal societies advocate informed dialysis selection and greater use of HoD to facilitate improvements in Veterans' post-ESRD clinical and health services utilization outcomes.

Reports from Europe and Canada show that providing comprehensive pre-ESRD patient education (CPE) improves the quality of CKD care and empowers patients to make informed dialysis modality selection. Data further show that informed modality selection substantially corrects the underuse of HoD as desired by the healthcare systems, including VHA.

However, across VHA, many Veterans with CKD are identified too late to benefit from CPE; and even for those identified and under renal care, the availability of CPE is limited. This results in suboptimal pre-ESRD care and preparation, and continued low HoD utilization. Thus, there is an urgent systemic need to provide CPE to all pre-ESRD (stage 4 and 5 CKD) Veterans and study its effectiveness prospectively within the VHA.

This study aims to evaluate the impact of the comprehensive pre-ESRD patient education on high-impact outcomes for Veterans and health services, across a local Veterans Healthcare System (VHS). The investigators will compare the impact of CPE (intervention), delivered either in-person or through telemedicine, with the usual care (control) enhanced by the provision of the self-learning CKD information among Veterans with advanced CKD across the North Florida/South Georgia VHS.

The investigators' study has four aims, consisting of one primary outcome (HoD use) and multiple secondary outcomes, to help us understand the impact of CPE on patients' informed decision making and on important post-ESRD clinical, patient-reported, and health services outcomes.

Aim 1: Compare the impact of CPE on Veterans' knowledge of CKD, their confidence in dialysis decision making, and their selection of dialysis modality, between the CPE and usual care groups.

H1.1: CPE will improve Veterans' knowledge of CKD and its management. H1.2: CPE will improve Veterans' confidence in making an informed selection of a dialysis modality.

H1.3: CPE will increase Veterans' selection of HoD. Aim 2: Compare Veterans' actual use of HoD (Primary Outcome) between the CPE and usual care groups.

H2.1: Veterans in the CPE group will show increased HoD use. Aim 3: Examine Veterans' perceived satisfaction with CPE, explore their preferences for F2F- or Tele-CPE, and investigate barriers and facilitators in the selection and use of their preferred dialysis modality. (Qualitative) Aim 4: Compare the following post-ESRD secondary outcomes between the CPE and usual care groups.

Patient reported outcomes: 1) health-related quality of life and 2) satisfaction with dialysis; clinical outcomes: 3) time to ESRD, 4) estimated glomerular filtration rate at ESRD, 5) need for inpatient initiation of dialysis, and 6) vascular access status at ESRD; and health services utilization outcomes: 7) number of inpatient stays, and 8) number of outpatient visits, from enrollment to 90-day post ESRD period.

H4: Veterans in the CPE group will show improvement in these secondary outcomes.

Findings from this study will help to achieve the long-term goal of better meeting the needs of Veterans with advanced CKD by improving Veterans' knowledge of CKD and its management, and promoting evidence-based Veteran-centered ESRD care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans registered to receive healthcare from the NF/SG VHS
* 18 years or older
* Advanced CKD (stage 4 or 5) and not on dialysis

Exclusion Criteria:

* Non-English speakers
* Veterans who are homeless or living in assisted living facilities or nursing homes
* Veterans with diagnosed dementia
* Veterans with the life-expectancy less than 6 months
* Any additional special concerns of a Veteran's provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Home Dialysis Use | 0-48 months
  Patient receiving either CPE or Enhanced usual care (EUC) will be followed for the diagnosis of ESRD and initiation of dialysis. The investigators will follow the use of peritoneal dialysis or home hemodialysis at day 90 into the dialysis as the home dialysis (HoD) use primary outcome.

SECONDARY OUTCOMES:
Home Dialysis selection | 0-4 weeks
  post-CPE/EUC dialysis modality selection and examining the rates of home dialysis selection. post-CPE assessments will be made when subject is deemed confident in dialysis selection (see selection outcome). Post-EUC assessments will be made 10 days after the provision of the education material.
Kidney Disease Knowledge | 0-4 weeks
  pre- and post- kidney disease knowledge assessments after CPE/EUC. post-CPE assessments will be made when subject is deemed confident in dialysis selection (see selection outcome). Post-EUC assessments will be made 10 days after the provision of the education material.
confidence in dialysis decision making | 0-4 weeks
  post-CPE/EUC confidence in dialysis decision making. ). Intent-to-Teach will be assessed by confidence for dialysis decision making (defined by confidence rating of "quite confident" or "very confident"); those with suboptimal scores ("not at all confident" or "a little confident") or "uncertain of the dialysis modality choice," will undergo repeat CPE sessions weekly for up to 3 sessions. Based on our pilot studies showing the need for about 1.7 CPE session, the investigators expect that patients enrolled in CPE group will do post-CPE Aim 1 data collection (secondary outcome) at an average of 10 days
post-ESRD Kidney Disease Quality of life-36 | 3-48 months
  post CPE/EUC. This will only be measured in subjects that start dialysis therapy, 90 days post initiation of dialysis.
Satisfaction on Dialysis | 3-48 months
  post CPE/EUC. This will only be measured in subjects that start dialysis therapy, 90 days post initiation of dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh M. Shukla, MD MBBS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shukla AM, Cavanaugh KL, Jia H, Hale-Gallardo J, Wadhwa A, Fischer MJ, Reule S, Palevsky PM, Fried LF, Crowley ST. Needs and Considerations for Standardization of Kidney Disease Education in Patients with Advanced CKD. Clin J Am Soc Nephrol. 2023 Sep 1;18(9):1234-1243. doi: 10.2215/CJN.0000000000000170. Epub 2023 May 8. PMID 37150877
- [Result] Campbell-Montalvo R, Ftouni D, Shell P, Subhash S, Pearce K, Shukla AM. Understanding how patient education affects the process of treatment decision-making: Cultural model change in kidney disease therapy. Patient Educ Couns. 2025 Oct;139:109254. doi: 10.1016/j.pec.2025.109254. Epub 2025 Jul 5. PMID 40663840
- [Result] Pearce KE, Guo Y, Subhash S, Ftouni D, Visconti B, Wadhwa A, Agarwal A, Jia H, Shukla AM. Decision Readiness and Determinants of KRT among Veterans with Advanced CKD. Clin J Am Soc Nephrol. 2025 Apr 11;20(7):931-939. doi: 10.2215/CJN.0000000713. PMID 40215111
- [Result] Shukla AM, Visconti B, Pearce K, Orozco T, Hale-Gallardo J, Subhash S, Freytes IM, Jia H, Romero S, Guo Y. Development and Validation of KRT Knowledge Instrument. Clin J Am Soc Nephrol. 2024 Jul 1;19(7):877-886. doi: 10.2215/CJN.0000000000000472. Epub 2024 May 15. PMID 38748976
- [Result] Chamarthi G, Orozco T, Hale-Gallardo J, Subhash S, Shell P, Pearce K, Jia H, Shukla AM. Informed Dialysis Modality Selection Among Veterans With Advanced CKD: A Community-Level Needs Assessment. Kidney Med. 2024 Apr 26;6(6):100832. doi: 10.1016/j.xkme.2024.100832. eCollection 2024 Jun. PMID 38873241
- [Result] Chamarthi G, Orozco T, Shell P, Fu D, Hale-Gallardo J, Jia H, Shukla AM. Electronic Phenotype for Advanced Chronic Kidney Disease in a Veteran Health Care System Clinical Database: Systems-Based Strategy for Model Development and Evaluation. Interact J Med Res. 2023 Jul 24;12:e43384. doi: 10.2196/43384. PMID 37486757
- [Result] Campbell-Montalvo R, Jia H, Shukla AM. Supporting Shared Decision-Making and Home Dialysis in End-Stage Kidney Disease. Int J Nephrol Renovasc Dis. 2022 Sep 8;15:229-237. doi: 10.2147/IJNRD.S375347. eCollection 2022. PMID 36105650
- [Result] Orozco T, Segal E, Hinkamp C, Olaoye O, Shell P, Shukla AM. Development and validation of an end stage kidney disease awareness survey: Item difficulty and discrimination indices. PLoS One. 2022 Sep 9;17(9):e0269488. doi: 10.1371/journal.pone.0269488. eCollection 2022. PMID 36083893
- [Result] Shukla AM, Hale-Gallardo J, Orozco T, Freytes I, Purvis Z, Romero S, Jia H. A randomized controlled trial to evaluate and assess the effect of comprehensive pre-end stage kidney disease education on home dialysis use in veterans, rationale and design. BMC Nephrol. 2022 Mar 30;23(1):121. doi: 10.1186/s12882-022-02740-8. PMID 35354430
- [Result] Shukla AM, Cavanaugh KL, Wadhwa A, Crowley ST, Fried L. Basic Requirements for Improving Home Dialysis Utilization: Universal Access to Specialty Nephrology Care and Comprehensive Pre-ESKD Education. J Am Soc Nephrol. 2023 Jan 1;34(1):21-25. doi: 10.1681/ASN.2022060685. Epub 2022 Oct 25. No abstract available. PMID 36283810
- [Derived] Cheng XBJ, Chan CT. Systems Innovations to Increase Home Dialysis Utilization. Clin J Am Soc Nephrol. 2024 Jan 1;19(1):108-114. doi: 10.2215/CJN.0000000000000298. Epub 2023 Aug 31. PMID 37651291

DOCUMENTS (1):
  • Informed Consent Form (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04064086/ICF_000.pdf